CLINICAL TRIAL: NCT03636256
Title: Phase 1/2 Trial Evaluating the Safety and Tolerability of NanoDoce® Injection and Intravesical Instillation in Subjects With Urothelial Carcinoma
Brief Title: Evaluation of NanoDoce® in Participants With Urothelial Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NANODOCE-2017-02
Expanded Access: NCT04060628 (No longer available)
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urinary Bladder Neoplasm; Urinary Bladder Cancer; Urogenital Neoplasms; Urologic Neoplasms; Urologic Cancer; Malignant Tumor of the Urinary Bladder; Cancer of the Bladder
Keywords: non-muscle invasive bladder cancer; muscle invasive bladder cancer; high-risk bladder cancer; BCG-unresponsive bladder cancer; BCG failure; BCG-refractory bladder cancer; BCG-resistant bladder cancer; NMIBC; MIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Urogenital Neoplasms; Urologic Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Docetaxel; Administration, Intravesical; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Open-label, dose rising trial consisting of a dose escalation phase and a dose confirmation phase for direct injection doses. In the dose escalation phase, subjects will be enrolled in sequential cohorts of three subjects starting at the lowest concentration. The dose determined to be most suitable for further evaluation will enroll additional subjects to total up to 12 subjects at that dose level.
  The study will also dose escalate Groups 1 and 2 for the intravesical instillation of NanoDoce concentrations (2.0 and 3.0 mg/mL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-Muscle Invasive Bladder Cancer (Experimental): Subjects will be enrolled in sequential, dose escalating cohorts of NanoDoce direct injection (0.75, 1.5, 2.5, or 3.75 mg/mL). Subjects will also receive an initial NanoDoce intravesical instillation at 2.0 or 3.0 mg/mL and additional Induction (6 weekly NanoDoce intravesical instillations, followed by 6 weeks of rest) and Maintenance (3 weekly NanoDoce intravesical instillations, followed by 9 weeks of rest) instillations at 2.0 or 3.0 mg/mL.
  Interventions: Drug: NanoDoce (direct injection); Drug: NanoDoce (intravesical instillation) - Visit 2 Instillation; Drug: NanoDoce (intravesical instillation) - Induction and Maintenance Instillations
- Muscle Invasive Bladder Cancer (Experimental): Subjects will be enrolled in sequential, dose escalating cohorts of NanoDoce direct injection (0.75, 1.5, 2.5, or 3.75 mg/mL). Subjects will also receive an initial NanoDoce intravesical instillation at 2.0 or 3.0 mg/mL. Subjects will then go on to receive institutional standard of care.
  Interventions: Drug: NanoDoce (direct injection); Drug: NanoDoce (intravesical instillation) - Visit 2 Instillation; Other: Institutional Standard of Care

INTERVENTIONS:
Drug: NanoDoce (direct injection) — Subjects will receive NanoDoce injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT)
  Other Names: docetaxel; large surface area microparticle docetaxel
Drug: NanoDoce (intravesical instillation) - Visit 2 Instillation — All subjects will receive an initial intravesical instillation within 2 hours of direct injection.
  Other Names: docetaxel; large surface area microparticle docetaxel
Other: Institutional Standard of Care — Group 2 (MIBC) will receive institutional standard of care treatments after the Visit 2 intravesical instillation.
  Arms: Muscle Invasive Bladder Cancer
Drug: NanoDoce (intravesical instillation) - Induction and Maintenance Instillations — Group 1 (NMIBC) will receive intravesical instillations in an Induction Period and a Maintenance Period.
  Other Names: docetaxel; large surface area microparticle docetaxel
  Arms: Non-Muscle Invasive Bladder Cancer

SUMMARY:
This is a clinical trial studying the administration of NanoDoce as a direct injection to the bladder wall immediately after tumor resection and as an intravesical instillation. All participants will receive NanoDoce, and will be evaluated for safety and tolerability, as well as the potential effects of NanoDoce on urothelial carcinoma.

DETAILED DESCRIPTION:
In this clinical trial, subjects with high-risk non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancer (MIBC), will receive NanoDoce. Subjects will be stratified into two treatment groups, Group 1 (NMIBC) and Group 2 (MIBC). All subjects will receive NanoDoce injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT), followed by an initial NanoDoce intravesical instillation.

Once the TURBT resection site is healed (approximately 1 month), Group 1 (NMIBC) subjects will proceed to a 3-month Induction period (6 weekly NanoDoce intravesical instillations, followed by 6 weeks of rest). After the Induction period, following confirmation of non-recurrence, Group 1 subjects will proceed to a 3-month Maintenance period (3 weekly NanoDoce intravesical instillations, followed by 9 weeks of rest).

After NanoDoce direct injection and the initial intravesical instillation, Group 2 subjects will proceed to institutional standard of care and will not receive Induction or Maintenance intravesical instillations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18 years;
* Patients with either:

  * High-risk Non-Muscle Invasive Bladder Cancer (NMIBC);
  * Muscle Invasive Bladder Cancer (MIBC);
* Urothelial carcinoma confirmed by biopsy, urine cytology, computed tomography scan (CT) or other institution-approved diagnostic methodology;
* All visible tumors removed during bladder resection (TURBT);
* Performance Status (ECOG) 0-2 at study entry;
* Life expectancy of at least 6 months;
* Adequate marrow, liver, and renal function;

  * ANC ≥ 1.5 x 10^9/L;
  * Hemoglobin ≥ 9.5 grams/dL;
  * Platelets ≥ 75 x 10^9/L;
  * Total bilirubin ≤ 1.5x institutional ULN;
  * AST/ ALT ≤ 2.5x institutional ULN;
  * Creatinine ≤ 1.5x institutional ULN;
* Adequate method of birth control.

Exclusion Criteria:

* Metastatic disease;
* Previous (within 12 months) or concurrent history of non-bladder malignancy, except for non-melanoma skin cancer;
* Intravesical therapy within 6 weeks prior to consent (chemotherapy or immunotherapy including BCG administered directly into the bladder);
* Resection surface area greater than 8 cm2;
* Upper tract and urethral disease within 18 months;
* Known hypersensitivity to any of the study drug components or reconstitution components;
* Pregnant or breastfeeding;
* Participation in the treatment phase of another clinical trial within 3 months prior to consent;
* Investigator's opinion of subject's probable noncompliance or inability to understand the trial and/or give adequate informed consent;
* Ongoing drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lamm, MD, FACS, Principal Investigator — BCG Oncology, PC
Locations (5):
- United States (5):
  - BCG Oncology, PC, Phoenix, Arizona
  - James Buchanan Brady Urological Institute, Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 0.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 1.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 or 3.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL: NanoDoce (direct injection): Subject received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subject received an initial intravesical instillation of NanoDoce at 3.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subject received intravesical instillations of NanoDoce at 3.0 mg/mL in an Induction Period (6 weekly NanoDoce intravesical instillations, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 0.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 1.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 3.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
Period: Overall Study
Arm/Group | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL
Started | 4 | 3 | 3 | 9 | 1 | 5 | 2 | 2 | 7
Completed | 1 | 3 | 1 | 8 | 1 | 1 | 0 | 2 | 2
Not Completed | 3 | 0 | 2 | 1 | 0 | 4 | 2 | 0 | 5
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1 | 0 | 4 | 2 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL | Total
Number analyzed (Participants) | 4 | 3 | 3 | 9 | 1 | 5 | 2 | 2 | 7 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 4
  >=65 years | 4 | 2 | 3 | 7 | 1 | 5 | 2 | 2 | 6 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 2 | 8
  Male | 4 | 2 | 2 | 6 | 0 | 5 | 2 | 2 | 5 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 6
  Not Hispanic or Latino | 4 | 3 | 2 | 8 | 1 | 5 | 2 | 2 | 2 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  White | 4 | 3 | 3 | 8 | 1 | 4 | 2 | 2 | 6 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (Safety and Tolerability)
Description: Treatment Emergent Adverse Events included laboratory assessments, physical examination findings, and vital signs.
Time Frame: Up to End of Treatment (Month 6 for Group 1 and Group 2 Subset, and Day 45 for Group 2)
Measure: Count of Participants; unit: Participants
Groups:
- Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
Arm/Group | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL
Number analyzed (Participants) | 4 | 3 | 3 | 9 | 1 | 5 | 2 | 2 | 7
Participants | 3 | 3 | 3 | 9 | 1 | 5 | 2 | 1 | 6

2. Secondary Outcome: Recurrence Free Survival (RFS)
Description: No evidence of tumor recurrence or disease progression
Time Frame: At Months 6, 9, and 12
Population: All subjects from the NMIBC Group 1 were evaluated for RFS. No subjects in the MIBC Group 2 or MIBC Group 2 Subset were evaluated for RFS.
Measure: Mean (Standard Deviation); unit: Months
Groups:
- Non-Muscle Invasive Bladder Cancer - 0.75 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 0.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer - 1.5 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 1.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer - 2.5 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer - 3.75 NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 or 3.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
Arm/Group | Non-Muscle Invasive Bladder Cancer - 0.75 mg/mL NanoDoce Injection Cohort | Non-Muscle Invasive Bladder Cancer - 1.5 mg/mL NanoDoce Injection Cohort | Non-Muscle Invasive Bladder Cancer - 2.5 mg/mL NanoDoce Injection Cohort | Non-Muscle Invasive Bladder Cancer - 3.75 NanoDoce Injection Cohort
Number analyzed (Participants) | 4 | 3 | 3 | 9
Months | 5.1 (1.79) | 6.7 (3.10) | 4.7 (1.10) | 9.6 (3.31)

3. Secondary Outcome: Disease Progression
Description: Disease progression at Day 45 derived from cytology and biopsy assessments
Time Frame: Day 45
Population: The muscle invasive bladder cancer (MIBC) (Group 2) and MIBC Group 2 Subset were assessed for disease progression at Day 45. There were two subjects in the 3.75 mg/mL NanoDoce cohort for whom disease status at Day 45 was unknown, and there were two subjects withdrawn from the study prior to analysis of disease progression at Day 45.
Measure: Count of Participants; unit: Participants
Groups:
- Muscle Invasive Bladder Cancer - 0.75 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 0.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer - 1.5 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 1.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer - 2.5 mg/mL NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 2.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL.
- Muscle Invasive Bladder Cancer - 3.75 NanoDoce Injection Cohort: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an intravesical instillation of NanoDoce 3.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Muscle Invasive Bladder Cancer Subset (Group 2 Subset) - 3.75/mg/mL NanoDoce Injection: NanoDoce (direct injection): Subject received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subject received an initial intravesical instillation of NanoDoce at 3.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subject received intravesical instillations of NanoDoce at 3.0 mg/mL in an Induction Period (6 weekly NanoDoce intravesical instillations, followed by 6 weeks of rest) and a Maintenance Period (3 weekly NanoDoce intravesical instillations, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
Arm/Group | Muscle Invasive Bladder Cancer - 0.75 mg/mL NanoDoce Injection Cohort | Muscle Invasive Bladder Cancer - 1.5 mg/mL NanoDoce Injection Cohort | Muscle Invasive Bladder Cancer - 2.5 mg/mL NanoDoce Injection Cohort | Muscle Invasive Bladder Cancer - 3.75 NanoDoce Injection Cohort | Muscle Invasive Bladder Cancer Subset (Group 2 Subset) - 3.75/mg/mL NanoDoce Injection
Number analyzed (Participants) | 5 | 2 | 2 | 3 | 1
Participants | 2 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: AE were captured from first study drug dose (injection) until 45 days after the last study drug dose (injection or instillation) for Group 2 subjects or until the End of Treatment (Visit 13 - Day 180) visit for Group 1 or Group 2 subset subjects. Subjects were required to spontaneously report any AEs. Study personnel asked open-ended questions to obtain information about AEs at every visit.
Description: Subjects were required to spontaneously report any AEs. Study personnel asked open-ended questions to obtain information about AEs at every visit.
Groups:
- Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 2.5 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 mg/mL or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period Maintenance (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation) - Subjects received an initial intravesical instillation of NanoDoce at 2.0 or 3.0 mg/mL within 2 hours of direct injection.
  NanoDoce (intravesical instillation) - Induction and Maintenance Instillations: Subjects received intravesical instillations of NanoDoce in an Induction Period (6 weekly NanoDoce intravesical instillations at 2.0 or 3.0 mg/mL, followed by 6 weeks of rest) and a Maintenance Period Maintenance (3 weekly NanoDoce intravesical instillations at 3.0 mg/mL, followed by 9 weeks of rest). Total dose administered for intravesical instillations could not exceed 50 mg in 25 mL of saline for a final concentration of 2.0 mg/mL or 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
- Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL: NanoDoce (direct injection): Subjects received NanoDoce 3.75 mg/mL (up to 4 mL) injected into the index tumor resection site on the bladder wall, immediately following transurethral resection of the bladder tumor (TURBT).
  NanoDoce (intravesical instillation): Subjects received an initial intravesical instillation of NanoDoce 3.0 mg/mL within 2 hours of direct injection. Total dose administered for intravesical instillation could not exceed 75 mg in 25 mL of saline for a final concentration of 3.0 mg/mL.
Arm/Group | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/9 | 0/1 | 0/5 | 0/2 | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 1/9 | 0/1 | 1/5 | 0/2 | 0/2 | 1/7
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 3/3 | 9/9 | 1/1 | 4/5 | 2/2 | 2/2 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL (N=4) | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL (N=3) | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL (N=3) | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL (N=9) | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL (N=1) | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL (N=5) | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL (N=2) | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL (N=2) | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL (N=7)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Kidney stone
Bladder Perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Muscle Invasive Bladder Cancer (Group 1) 0.75 mg/mL (N=4) | Non-Muscle Invasive Bladder Cancer (Group 1) 1.5 mg/mL (N=3) | Non-Muscle Invasive Bladder Cancer (Group 1) 2.5 mg/mL (N=3) | Non-Muscle Invasive Bladder Cancer (Group 1) 3.75 mg/mL (N=9) | Muscle Invasive Bladder Cancer (Group 2) Subset 3.75 mg/mL (N=1) | Muscle Invasive Bladder Cancer (Group 2) 0.75 mg/mL (N=5) | Muscle Invasive Bladder Cancer (Group 2) 1.5 mg/mL (N=2) | Muscle Invasive Bladder Cancer (Group 2) 2.5 mg/mL (N=2) | Muscle Invasive Bladder Cancer (Group 2) 3.75 mg/mL (N=7)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue Discoloration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corona Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Culture urine positive (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (6) | 1 (3) | 2 (3) | 3 (5) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urine abnormality (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT03636256/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/56/NCT03636256/SAP_001.pdf